CLINICAL TRIAL: NCT05341232
Title: A Lego Robot Programming Intervention for Enhancing Older Adult Cognitive Health
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Taiwan University Hospital (Other)
Collaborators: Ministry of Science and Technology, Taiwan (Other Government); National Taiwan University (Other); National Taiwan Science Education Center (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Basic Science
Other Study IDs: 202103148RINC
Record Dates: First submitted 2022-04-06; First posted 2022-04-22 (Actual); Last update posted 2026-02-05 (Actual); Status verified 2025-07

CONDITIONS: Cognitive Inferential Ability
Keywords: Aging; Cognitive Training Intervention; Lego Robot; Clinical Trial; Public Education; Psychological Testing; Brain Imaging

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Problem-Solving Training (Experimental): Participants will learn to program LEGO robots and will be encouraged to actively solve problems.
  Interventions: Behavioral: Lego Robot Programming Active Challenges; Behavioral: Lego Robot Programming Procedural Methods
- Step-By-Step Training (Active Comparator): Participants will learn to program LEGO robots and will be instructed step by step.
  Interventions: Behavioral: Lego Robot Programming Procedural Methods
- Board Games (Placebo Comparator): Participants will play boards games under a schedule matching the Experimental and Active Comparator arms.
  Interventions: Behavioral: Board Games

INTERVENTIONS:
Behavioral: Lego Robot Programming Active Challenges — Participants will adapt their own Lego robot programs to achieve specific task goals.
  Arms: Problem-Solving Training
Behavioral: Lego Robot Programming Procedural Methods — Participating will undergo Lego robot programming training that engages them to follow fixed programming coding steps.
  Arms: Problem-Solving Training; Step-By-Step Training
Behavioral: Board Games — Participants will play board games with each other.
  Arms: Board Games

SUMMARY:
The population in Taiwan is rapidly aging with an increasing proportion of older persons who experience cognitive difficulties but are otherwise physically healthy. As such there is a critical and urgent need for effective interventions to enhance older adult cognitive health. This present sub-project is part of the larger integrated project that will address this need by conducting cognitive training interventions on community older adults using the National Taiwan Science Education Center (NTSEC) as the public engagement window and collecting research behavioral and neurophysiological data to empirically and objectively examine intervention efficacies. In this sub-project, the investigators implement a clinical trial to evaluate an open-ended, flexible cognitive training intervention in middle to older adults aged 50 yrs or above using a 12-week Lego Robot Programming (Lego RP) protocol developed in the investigators' lab at the Graduate Institute of Brain and Mind Sciences, College of Medicine, National Taiwan University. The Lego RP training requires participants to generate and update abstract mental hypotheses of the effect of program codes on the physical actions of a robot based on how the robot behaves. Such mental processing is thought to drive flexible coordination between neural processes in the brain and benefit a broad range of cognitive abilities in older adults. The investigators target to obtain pre- and post-intervention behavioral and neurophysiological data (including brain imaging indicators) in 40 experimental participants, 40 active control participants, and 40 passive control participants over a period of 3 years.

DETAILED DESCRIPTION:
The population in Taiwan is rapidly aging with an increasing proportion of older persons who experience cognitive difficulties but are otherwise physically healthy. As such there is a critical and urgent need for effective interventions to enhance older adult cognitive health. This present sub-project is part of the larger integrated project that will address this need by conducting cognitive training interventions on community older adults using the National Taiwan Science Education Center (NTSEC) as the public engagement window and collecting research behavioral and neurophysiological data to empirically and objectively examine intervention efficacies. In this sub-project, the investigators implement a clinical trial to evaluate an open-ended, flexible cognitive training intervention in middle to older adults aged 50 yrs or above using a 12-week Lego Robot Programming (Lego RP) protocol developed in the investigators' lab at the Graduate Institute of Brain and Mind Sciences, College of Medicine, National Taiwan University. The Lego RP training requires participants to generate and update abstract mental hypotheses of the effect of program codes on the physical actions of a robot based on how the robot behaves. Such mental processing is thought to drive flexible coordination between neural processes in the brain and benefit a broad range of cognitive abilities in older adults. The investigators target to obtain pre- and post-intervention behavioral and neurophysiological data (including brain imaging indicators) in 40 experimental participants, 40 active control participants, and 40 passive control participants over a period of 3 years. The investigators will also coordinate with the other sub-projects to assign participants to the different interventions involved as well as research data collection, which is shared. In contrast to previous studies of older adult cognitive training, the investigators expect this present approach, which leverages neurocognitive principles, to result in notable transfer between different cognitive abilities, and meaningful impact on daily functioning. The NTSEC recently seeks to engage the public, particularly children and older adults in STEAM education (Science, Technology, Engineering, Arts, Mathematics) to inspire and equip the population with the spirit of learning, discovery, and challenge-seeking, which is thought to raise mental resilience. Thus, the investigators' public outreach and research goals are highly complementary and the work is expected to yield more ecologically valid research data on a novel class of cognitive interventions for cognitive aging using psychological and brain imaging techniques to bridge critical neural mechanistic knowledge gaps. In addition, the research study will apply real public education benefits in society for those approximately 300 older participants who will participate in this study.

ELIGIBILITY:
Inclusion Criteria:

* Literate in Mandarin and Taiwanese
* Willing and able to participate in this research protocol in its entirety.
* Age >65

Exclusion Criteria:

* Participated in cognitive-related training in the past two months.
* Diagnosed with mild cognitive impairment (MCI)
* Severe psychological or behavioral disorder that would seriously interfere with the progress of activity
* History of degenerative cognitive disorder.
* Counter-indications for MRI scanning.

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 48 (Actual)
Dates: Start 2021-09-01 (Actual); Primary Completion 2025-03-20 (Actual); Study Completion 2025-03-20 (Actual)

PRIMARY OUTCOMES:
Changes of neural functional activity during inferential processing | Week 0, Week 12
  Participants will undergo a Rule Inference fMRI task to infer underlying rules that map color configurations of circles in a triangular arrangement to a target color category within as few tries as possible under active or passive conditions. The goal for participants will be to infer the cue-category association rules using as few cues as possible. The primary outcome measure here is the degree of neural response estimate change in blood oxygen level dependent (BOLD) signal pre- and post-intervention.
Changes of overall accuracy during inferential processing | Week 0, Week 12
  Changes from pre- to post-intervention in participant overall accuracy in identifying latent rules in the Rule Inference fMRI task.
Changes of learning rate during inferential processing | Week 0, Week 12
  Changes from pre- to post-intervention in participant number of trials to criterion in the Rule Inference fMRI task.
Changes of strategic performance during inferential processing | Week 0, Week 12
  Changes from pre- to post-intervention in participant coefficients of expression of modeled response strategies in the Rule Inference fMRI task will be assessed.
Changes in the Montreal Cognitive Assessment (MoCA) score | Week 0, Week 12
  Pre- to post-intervention changes in participant MoCA score. Score range from 0 to 30 with higher scores indicating better cognitive ability.
Change in Wechsler Memory Scale III Logical Memory I & II | Week 0, Week 12
  Score range 0 - 75. Higher score indicates better verbal episodic memory.
Change in Wechsler Memory Scale III Face Memory | Week 0, Week 12
  Score range 0 - 48. Higher score indicates better visual face memory.
Change in Wechsler Memory Scale III Verbal Paired Memory | Week 0, Week 12
  Score range 0 - 32. Higher score indicates better verbal memory and learning.
Change in Wechsler Memory Scale III Family Pictures I & II | Week 0, Week 12
  Score range 0 - 64. Higher score indicates better visual memory and learning.
Change in Wechsler Memory Scale III Word Lists I & II | Week 0, Week 12
  Score range 0 - 36. Higher score indicates better verbal memory and learning. For II, recall score range is 0 to 8; recognition score range is 0 to 24.
Change in Wechsler Memory Scale III Visual Reproduction I & II | Week 0, Week 12
  Score range 0 - 104. Higher score indicates better visual memory. For II, recall score range is 0-104; recognition score range is 0-48.
Change in Wechsler Memory Scale III Spatial Span | Week 0, Week 12
  Score range 0 - 32. Higher score indicates better spatial memory.
Change in Wechsler Memory Scale III Digit Span | Week 0, Week 12
  Score range 0 - 32. Higher score indicates better auditory memory.
Change in Wechsler Adult Intelligence Scale III Vocabulary | Week 0, Week 12
  Score range 0 - 66. Higher score indicates better vocabulary.
Change in Wechsler Adult Intelligence Scale III Digit Symbol | Week 0, Week 12
  Score range 0 - 133. Higher score indicates better processing speed.
Change in Wechsler Adult Intelligence Scale III Block Design | Week 0, Week 12
  Score range 0 - 68. Higher score indicates better visual processing.
Change in Wechsler Adult Intelligence Scale III Arithmetic | Week 0, Week 12
  Score range 0 - 22. Higher score indicates better mathematical computation ability.
Change in Wechsler Adult Intelligence Scale III Matrix Reasoning | Week 0, Week 12
  Score range 0 - 26. Higher score indicates better reasoning.

SECONDARY OUTCOMES:
Changes of neural functional activity during resting-state | Week 0, Week 12
  Brain functional activity measured using fMRI during rest with eyes-open.

CONTACTS AND LOCATIONS:
Overall Officials: Joshua OS Goh, Ph. D., Principal Investigator — National Taiwan University
Locations (2):
- Taiwan (2):
  - College of Medicine, National Taiwan University, Taipei
  - National Taiwan Science Education Center, Taipei

IPD SHARING:
Plan to Share IPD: Yes
Data that can be shared include anonymized neuropsychological assessment scores, cognitive behavioral performance scores, brain imaging data that have been published.
Supporting Information: Study Protocol, SAP, Analytic Code
Time Frame: Data will become available 1 year after primary results are published by the central research team. Data are anticipated to be available for sharing for an indefinite period after the above criteria is met.
Access Criteria: Data sharing will be done based direct requests and on case-by-case evaluation for appropriateness. Use of shared data will require agreement on appropriate citation of data sources at least or authorship inclusion or acknowledgement.